CLINICAL TRIAL: NCT00946283
Title: Probiotic Enteric Regimen For Easing Complications of Transplant : A Pilot Study (PERFECT Trial)
Brief Title: Lactobacillus in Preventing Infection in Patients Undergoing a Donor Stem Cell Transplant for Hematologic Cancer or Myelodysplastic Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 060802; P30CA072720 (NIH); CDR0000649274 (Other: NIH); 0220090096 (Other: IRB); NCI-2012-00597 (Other: NCI)
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Breast Cancer; Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Neuroblastoma; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent mycosis fungoides/Sezary syndrome; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent malignant testicular germ cell tumor; secondary myelodysplastic syndromes; stage II multiple myeloma; stage III multiple myeloma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; refractory multiple myeloma
MeSH Terms: conditions — Breast Neoplasms; Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neuroblastoma; Ovarian Neoplasms; Testicular Germ Cell Tumor; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Acute; Leukemia, Hairy Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Carcinoma, Ovarian Epithelial; Testicular Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lactobacillus GG (Experimental): Open label trial of Culturelle (Lactobacillus GG) administered to patients after engraftment, post allogeneic stem cell transplantation.
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus GG — Culturelle DS (Lactobacillus GG) will be administered one capsule (10 billion live lactobacillus GG) daily with water
  Other Names: Culturelle DS

SUMMARY:
RATIONALE: Probiotics, such as Lactobacillus, may be effective in preventing infections in patients with suppressed immune systems.

PURPOSE: This phase I trial is studying the side effects and how well giving enteral nutrition, including Lactobacillus, works in preventing infections in patients undergoing donor stem cell transplant for hematologic cancer or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if patients who are treated with a probiotic-containing diet develop infection with one of the probiotic microorganisms while undergoing allogenic hematopoietic stem cell transplantation for a hematologic malignancy or myelodysplastic syndrome.

OUTLINE: Patients receive oral Lactobacillus rhamosus GG (Culturelle DS) once daily beginning when blood counts have recovered without filgrastim (G-CSF) or sargramostim (GM-CSF) support for 3 consecutive days and continuing for 1 year after transplantation.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Currently undergoing allogeneic stem cell transplantation from a related or unrelated donor for a hematologic malignancy or myelodysplastic syndrome
* Hematopoietic engraftment as evidenced by recovery of the absolute neutrophil count > 1000/μL for > 3 days without filgrastim (G-CSF) support within 30 days of transplant

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Serum creatinine ≤ 2.0
* AST or ALT ≤ 3 times upper limit of normal (ULN)
* Total bilirubin ≤ 2.0 times ULN
* No clostridium difficile enterocolitis diagnosed during the transplant hospitalization in the peri-transplant period
* Able to take medications by mouth
* No evidence of graft-vs-host disease
* No history of inflammatory bowel disease or other chronic diarrheal illness
* No history of hypersensitivity to milk proteins

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 months since prior use of probiotics supplements, excluding yogurt and cheeses with live cultures
* No concurrent over-the-counter medications or herbal remedies

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2013-05 (Actual); Study Completion 2015-10-14 (Actual)

PRIMARY OUTCOMES:
Safety as indicated by the lack of infection attributable to probiotic organisms | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, MD, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States